CLINICAL TRIAL: NCT05095662
Title: Establish a Specific Cohort Database for Depressive Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai 10th People's Hospital (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHDC2020CR6023
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-04

CONDITIONS: Depressive Disorder
Keywords: depression; cohort study; database
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depression is characterized by high prevalence, high recurrence rate, high disability rate, high suicide rate, and heavy disease burden. However, the diagnosis, treatment, and prognosis of depression are difficult to meet the clinical needs at present. This study plans to integrate a large sample of hospital clinical data, laboratory examination data, brain imaging, and electrophysiological data, as well as audio-visual data, to establish a database for depressive disorder, and long-term follow-up to form a specific disease cohort. This study will provide a scientific basis for exploring biomarkers related to objective diagnosis and treatment of depression.

DETAILED DESCRIPTION:
Together with three tertiary hospitals in Shanghai, Shanghai Tenth People's Hospital, Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine, and Zhongshan Hospital affiliated to Fudan University, Shanghai Mental Health Center will take a lead to establish a big database focused on depressive disorders. Expert consensus will be used to determine the standard for the dataset. Real-world data will be include. To establish a depressive disorders-specific database with multiple functions, such as data insight, data retrieval, cohort project establishment, follow-up, and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Meeting ICD-10 depressive episode criteria (F32, F33, F34, F38, F39)
* Cultural, social and educational background sufficient to understand informed consent and research content
* Agree to participate in this study

Exclusion Criteria:

* Exclude other mental disorders such as bipolar disorder and schizophrenia (but not comorbidities)
* Patients with a history of brain injury or cerebrovascular accident, myocardial infarction, severe liver cirrhosis, acute and chronic renal failure, severe diabetes, aplastic anemia, moderate and severe malnutrition and other serious physical diseases of the nervous, heart, liver, kidney, endocrine and blood systems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Depressive disorder cohort study: Outpatient or inpatient patients in Shanghai Mental Health Center, Shanghai Zhongshan Hospital, Renji Hospital and Shanghai Tenth People's Hospital were included in this cohort study if the patients agreed to participate in this study and the patients with depressive disorder met the inclusion and exclusion criteria.
  2. Construction of standard database for depression: All inpatients and outpatients of Shanghai Mental Health Center will be included in the special database if they meet the diagnostic criteria for depression（ICD-10）.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Construct the structured data set for depression by integrating a large sample of outpatient and inpatient clinical data, blood tests, psychological tests, and brain imaging data. | 3 years
  Have 80000 patients been included.

SECONDARY OUTCOMES:
Recruitment of 300 patients who was diagnosed as depressive disorders. | Baseline, and 1,2,3,4,5 years follow-up point
  In order to: collect demographic and sociological information., clinical data, social function, cognitive function, and blood index test. Collection of Audio-Visual, as well as brain imaging or electrophysiology if patients agreed to participate in these tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, M.D., Ph.D., Principal Investigator — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips MR, Zhang J, Shi Q, Song Z, Ding Z, Pang S, Li X, Zhang Y, Wang Z. Prevalence, treatment, and associated disability of mental disorders in four provinces in China during 2001-05: an epidemiological survey. Lancet. 2009 Jun 13;373(9680):2041-53. doi: 10.1016/S0140-6736(09)60660-7. PMID 19524780
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Gunaratne P, Lloyd AR, Vollmer-Conna U. Mood disturbance after infection. Aust N Z J Psychiatry. 2013 Dec;47(12):1152-64. doi: 10.1177/0004867413503718. Epub 2013 Sep 20. PMID 24056922
- [Background] Reppermund S, Ising M, Lucae S, Zihl J. Cognitive impairment in unipolar depression is persistent and non-specific: further evidence for the final common pathway disorder hypothesis. Psychol Med. 2009 Apr;39(4):603-14. doi: 10.1017/S003329170800411X. Epub 2008 Jul 30. PMID 18667101
- [Background] Anoushiravani AA, Patton J, Sayeed Z, El-Othmani MM, Saleh KJ. Big Data, Big Research: Implementing Population Health-Based Research Models and Integrating Care to Reduce Cost and Improve Outcomes. Orthop Clin North Am. 2016 Oct;47(4):717-24. doi: 10.1016/j.ocl.2016.05.008. Epub 2016 Aug 8. PMID 27637658
- [Background] Murphy DR, Meyer AN, Bhise V, Russo E, Sittig DF, Wei L, Wu L, Singh H. Computerized Triggers of Big Data to Detect Delays in Follow-up of Chest Imaging Results. Chest. 2016 Sep;150(3):613-20. doi: 10.1016/j.chest.2016.05.001. Epub 2016 May 10. PMID 27178786
- [Background] Auffray C, Balling R, Barroso I, Bencze L, Benson M, Bergeron J, Bernal-Delgado E, Blomberg N, Bock C, Conesa A, Del Signore S, Delogne C, Devilee P, Di Meglio A, Eijkemans M, Flicek P, Graf N, Grimm V, Guchelaar HJ, Guo YK, Gut IG, Hanbury A, Hanif S, Hilgers RD, Honrado A, Hose DR, Houwing-Duistermaat J, Hubbard T, Janacek SH, Karanikas H, Kievits T, Kohler M, Kremer A, Lanfear J, Lengauer T, Maes E, Meert T, Muller W, Nickel D, Oledzki P, Pedersen B, Petkovic M, Pliakos K, Rattray M, I Mas JR, Schneider R, Sengstag T, Serra-Picamal X, Spek W, Vaas LA, van Batenburg O, Vandelaer M, Varnai P, Villoslada P, Vizcaino JA, Wubbe JP, Zanetti G. Making sense of big data in health research: Towards an EU action plan. Genome Med. 2016 Jun 23;8(1):71. doi: 10.1186/s13073-016-0323-y. PMID 27338147